CLINICAL TRIAL: NCT02697279
Title: Evaluation of Loop Drainage Technique Versus Standard Incision and Drainage for Treatment of Simple Soft Tissue Abscesses
Brief Title: Loop Drainage: Effectiveness in Treating Cutaneous Abscesses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll the appropriate number of subjects within a reasonable timeframe.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Richard Gentry Wilkerson, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00066974
Record Dates: First submitted 2016-02-04; First posted 2016-03-03 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Abscess of Skin and/or Subcutaneous Tissue
Keywords: Abscess; Loop; Drainage
MeSH Terms: conditions — Abscess | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Incision and Drainage (Active Comparator): Treatment of a simple cutaneous abscess with traditional incision and drainage with or without packing, decision made at the discretion of the provider.
  Interventions: Procedure: Traditional Incision and Drainage.
- Loop drainage (Experimental): Treatment of a simple cutaneous abscess with incision and drainage using the loop drainage technique.
  Interventions: Procedure: Loop drainage

INTERVENTIONS:
Procedure: Traditional Incision and Drainage. — Control Group- Standard treatment of a simple cutaneous abscess with traditional I&D technique with or without packing utilizing a standard I&D kit.
  Arms: Traditional Incision and Drainage
Procedure: Loop drainage — Study Group- Treatment of a simple cutaneous abscess with the loop drainage technique utilizing an standard I&D kit and the cuff of a sterile glove for a loop device.
  Arms: Loop drainage

SUMMARY:
In the Emergency Department (ED), patients frequently seek medical treatment for cutaneous abscesses. Traditional incision and drainage (I&D), with or without packing of cutaneous abscesses has long been the accepted standard of care. This procedure is often very painful for the patient. Additionally, compliance with wound care and follow-up can present barriers to proper care and healing. Research has suggested that incision and loop drainage of an abscess may be another effective treatment for simple cutaneous abscess. Thus far, research into this procedure has been limited to the pediatric population with small sample sizes. In these previous studies, this technique was found to be an effective and less painful treatment for abscesses. Research has not been done in the adult population using this procedure. If this procedure is found to be as effective and less painful in the adult population, then it should be considered as a potential preferred I&D method for cutaneous abscess in the ED.

DETAILED DESCRIPTION:
Patients who meet study criteria for treatment of a simple cutaneous abscess and desire to be a part of this study, will be consented. Study subjects will be enrolled and randomly assigned to either the study or control groups.

Control Group- standard I & D method for cutaneous abscess.

Study Group- Loop Technique:

1. Gather all of your material and bring to bedside
2. Clean area with chlorhexidine or iodine swabs
3. Anesthetize area
4. Use your scalpel to make small 5mm incision at most fluctuant area of abscess
5. Explore cavity with your hemostat and break down loculations
6. Make second incision less than 4cm away from first incision. Feel borders of abscess, and try to make second incision as far within cavity as you can.
7. For larger abscesses can repeat step 5 thus creating several LOOPs.
8. Irrigate cavity with saline flush
9. Pass hemostat through both incisions and pull loop vessel, penrose, or bottom of glove through. Keep your loop device equal in length on both sides.
10. Tie loop device loosely over 30cc syringe to form LOOP. Usually 5-6 knots. This helps prevent loop from falling out prematurely.
11. Slide syringe out, and trim free ends of loop. Make sure loop is mobile.
12. Cover site with dry dressing. Follow-Up-

    * Wound check in 1-2 days
    * Patient may manage drain at home by rotating it to facilitate drainage and prevent adhesion
    * Patient will be instructed to return to the Emergency Department for drain removal in 5-7 days.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Presents to ED with simple cutaneous abscess
3. Provides informed consent.

Exclusion Criteria:

1. Under 18 years of age
2. Abscess too small for performance of procedure
3. Signs of systemic infection
4. Need for hospitalization
5. Previously treated for current abscess
6. Clinician determines abscess would not be amenable to drainage by loop technique
7. Patients known to be pregnant
8. Incarcerated patients
9. Students / Employees of the facility
10. Presence of any other condition(s) that the investigator feels makes the patient unsuitable for study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Procedure failure rate | 5 -7 days after procedure
  Determining the difference in failure rates between the study group and control group. Treatment failure is a composite outcome defined as having the presence of any of the following: requiring a 2nd incision and drainage procedure, a patient that requires administration of antibiotics after the initial treatment period due to worsening clinical status, a patient that requires hospitalization after the initial treatment period due to worsening clinical status.

SECONDARY OUTCOMES:
Difference in pain associated with the procedure using a visual analog pain scale | Measured after the procedure on day 1
  To evaluate the difference in pain between the experimental and control groups associated with the procedure using a visual analog pain scale (0-100).
Patient Satisfaction using a visual analog pain scale | 5-7 days after procedure
  To measure the difference in patient satisfaction with overall treatment between the study and control groups using the visual analog scale (0-100).

CONTACTS AND LOCATIONS:
Overall Officials: R. Gentry Wilkerson, MD, Principal Investigator — U of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ladd AP, Levy MS, Quilty J. Minimally invasive technique in treatment of complex, subcutaneous abscesses in children. J Pediatr Surg. 2010 Jul;45(7):1562-6. doi: 10.1016/j.jpedsurg.2010.03.025. PMID 20638546
- [Background] Kushnir VA, Mosquera C. Novel technique for management of Bartholin gland cysts and abscesses. J Emerg Med. 2009 May;36(4):388-90. doi: 10.1016/j.jemermed.2008.05.019. Epub 2008 Nov 26. PMID 19038518
- [Background] Ladde JG, Baker S, Rodgers CN, Papa L. The LOOP technique: a novel incision and drainage technique in the treatment of skin abscesses in a pediatric ED. Am J Emerg Med. 2015 Feb;33(2):271-6. doi: 10.1016/j.ajem.2014.10.014. Epub 2014 Oct 16. PMID 25435407
- [Background] Thompson DO. Loop drainage of cutaneous abscesses using a modified sterile glove: a promising technique. J Emerg Med. 2014 Aug;47(2):188-91. doi: 10.1016/j.jemermed.2014.04.035. Epub 2014 Jun 11. PMID 24928539
- [Background] McNamara WF, Hartin CW Jr, Escobar MA, Yamout SZ, Lau ST, Lee YH. An alternative to open incision and drainage for community-acquired soft tissue abscesses in children. J Pediatr Surg. 2011 Mar;46(3):502-6. doi: 10.1016/j.jpedsurg.2010.08.019. PMID 21376200
- [Background] Tsoraides SS, Pearl RH, Stanfill AB, Wallace LJ, Vegunta RK. Incision and loop drainage: a minimally invasive technique for subcutaneous abscess management in children. J Pediatr Surg. 2010 Mar;45(3):606-9. doi: 10.1016/j.jpedsurg.2009.06.013. PMID 20223328
- [Background] Taira BR, Singer AJ, Thode HC Jr, Lee CC. National epidemiology of cutaneous abscesses: 1996 to 2005. Am J Emerg Med. 2009 Mar;27(3):289-92. doi: 10.1016/j.ajem.2008.02.027. PMID 19328372